CLINICAL TRIAL: NCT01300390
Title: Assessment of Endothelial Function, Apolipoproteins, and Adiponectin Levels as Markers of Cardiovascular Before and After Liver Transplantation
Brief Title: Assessment of Endothelial Function, Apolipoproteins and Adiponectin
Acronym: Endo-PAT
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kymberly D. Watt, M.D., Mayo Clinic
Other Study IDs: 10-008776
Record Dates: First submitted 2011-02-17; First posted 2011-02-21 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Cirrhosis
Keywords: liver transplant; end-stage liver disease; cirrhosis
MeSH Terms: conditions — Fibrosis; End Stage Liver Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples will be retained for future liver transplant research.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- End-stage liver disease pre-transplant: Patients with end-stage liver disease (non-fulminant) awaiting liver transplant

SUMMARY:
The overall hypothesis is that endothelial function, apolipoprotein levels and adiponectin levels are accurate predictors of underlying cardiovascular disease in patients with end-stage liver disease, in whom standard tools for the diagnosis of and screening for cardiovascular disease are of limited utility.

DETAILED DESCRIPTION:
This study is looking at using a noninvasive test called a reactive hyperemia peripheral artery tonometry (RH-PAT) to check endothelial dysfunction. Endothelial dysfunction is thought to be an indication of future heart disease or metabolic disorders. Adiponectin is a hormone associated with heart disease. Apolipoprotein levels, are established risk factors for coronary artery disease in the general population. Our group would like to see if there is a link between endothelial function, adiponectin, apolipoprotein levels and posttransplant heart disease complications. The study would be taking these results to find new clinical procedures for patients that are at potentially higher risk of heart problems during and after their liver transplant procedure.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 21 years of age.
* Cirrhotic end-stage liver disease
* Pre-transplant

Exclusion Criteria:

* Dialysis shunt
* non-cirrhotic liver disease
* fulminant hepatic failure

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhotic end-stage liver disease awaiting transplant
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2011-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Endothelial dysfunction in cirrhotic liver transplant candidates up to one year after transplant. | one year posttransplant
  Endothelial function testing will be performed by reactive hyperemia peripheral artery tonometry in consecutive patients ≥21 years old awaiting liver transplantation and repeated at 3 weeks, 4 months and 1 year post transplantation

SECONDARY OUTCOMES:
Metabolic abnormalities and cardiovascular disease by endothelial dysfunction and blood testing up to one year pre-transplant | 1 year posttransplant
  Endothelial dysfunction testing, apolipoproteins and adiponectin levels will be performed prior to liver transplantation and repeated at 3 weeks (endothelial dysfunction only), 4 months and 1 year post transplantation. Pre transplant results will be analyzed for association with perioperative cardiovascular events. In addition, post transplant endothelial dysfunction results (and the delta change) along with adiponectin levels will be analyzed for cardiovascular event endpoints by 1 year post transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Kymberly Watt, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Carey WD, Dumot JA, Pimentel RR, Barnes DS, Hobbs RE, Henderson JM, Vogt DP, Mayes JT, Westveer MK, Easley KA. The prevalence of coronary artery disease in liver transplant candidates over age 50. Transplantation. 1995 Mar 27;59(6):859-64. PMID 7701580
- [Background] Tiukinhoy-Laing SD, Rossi JS, Bayram M, De Luca L, Gafoor S, Blei A, Flamm S, Davidson CJ, Gheorghiade M. Cardiac hemodynamic and coronary angiographic characteristics of patients being evaluated for liver transplantation. Am J Cardiol. 2006 Jul 15;98(2):178-81. doi: 10.1016/j.amjcard.2006.01.089. Epub 2006 May 12. PMID 16828588
- [Background] Diedrich DA, Findlay JY, Harrison BA, Rosen CB. Influence of coronary artery disease on outcomes after liver transplantation. Transplant Proc. 2008 Dec;40(10):3554-7. doi: 10.1016/j.transproceed.2008.08.129. PMID 19100436
- [Background] John PR, Thuluvath PJ. Outcome of liver transplantation in patients with diabetes mellitus: a case-control study. Hepatology. 2001 Nov;34(5):889-95. doi: 10.1053/jhep.2001.29134. PMID 11679959
- [Background] Bianchi G, Marchesini G, Marzocchi R, Pinna AD, Zoli M. Metabolic syndrome in liver transplantation: relation to etiology and immunosuppression. Liver Transpl. 2008 Nov;14(11):1648-54. doi: 10.1002/lt.21588. PMID 18975273
- [Background] Reuben A. Long-term management of the liver transplant patient: diabetes, hyperlipidemia, and obesity. Liver Transpl. 2001 Nov;7(11 Suppl 1):S13-21. doi: 10.1053/jlts.2001.29167. PMID 11689772
- [Background] Leonard J, Heimbach JK, Malinchoc M, Watt K, Charlton M. The impact of obesity on long-term outcomes in liver transplant recipients-results of the NIDDK liver transplant database. Am J Transplant. 2008 Mar;8(3):667-72. doi: 10.1111/j.1600-6143.2007.02100.x. PMID 18294163
- [Background] Moller S, Henriksen JH. Cirrhotic cardiomyopathy: a pathophysiological review of circulatory dysfunction in liver disease. Heart. 2002 Jan;87(1):9-15. doi: 10.1136/heart.87.1.9. PMID 11751653
- [Background] Therapondos G, Flapan AD, Plevris JN, Hayes PC. Cardiac morbidity and mortality related to orthotopic liver transplantation. Liver Transpl. 2004 Dec;10(12):1441-53. doi: 10.1002/lt.20298. PMID 15558590
- [Background] Keeffe BG, Valantine H, Keeffe EB. Detection and treatment of coronary artery disease in liver transplant candidates. Liver Transpl. 2001 Sep;7(9):755-61. doi: 10.1053/jlts.2001.26063. PMID 11552207
- [Background] Findlay JY, Keegan MT, Pellikka PP, Rosen CB, Plevak DJ. Preoperative dobutamine stress echocardiography, intraoperative events, and intraoperative myocardial injury in liver transplantation. Transplant Proc. 2005 Jun;37(5):2209-13. doi: 10.1016/j.transproceed.2005.03.023. PMID 15964381
- [Background] Umphrey LG, Hurst RT, Eleid MF, Lee KS, Reuss CS, Hentz JG, Vargas HE, Appleton CP. Preoperative dobutamine stress echocardiographic findings and subsequent short-term adverse cardiac events after orthotopic liver transplantation. Liver Transpl. 2008 Jun;14(6):886-92. doi: 10.1002/lt.21495. PMID 18508373
- [Background] Takase B, Uehata A, Akima T, Nagai T, Nishioka T, Hamabe A, Satomura K, Ohsuzu F, Kurita A. Endothelium-dependent flow-mediated vasodilation in coronary and brachial arteries in suspected coronary artery disease. Am J Cardiol. 1998 Dec 15;82(12):1535-9, A7-8. doi: 10.1016/s0002-9149(98)00702-4. PMID 9874063
- [Background] Bonetti PO, Pumper GM, Higano ST, Holmes DR Jr, Kuvin JT, Lerman A. Noninvasive identification of patients with early coronary atherosclerosis by assessment of digital reactive hyperemia. J Am Coll Cardiol. 2004 Dec 7;44(11):2137-41. doi: 10.1016/j.jacc.2004.08.062. PMID 15582310
- [Background] Yeboah J, Crouse JR, Hsu FC, Burke GL, Herrington DM. Brachial flow-mediated dilation predicts incident cardiovascular events in older adults: the Cardiovascular Health Study. Circulation. 2007 May 8;115(18):2390-7. doi: 10.1161/CIRCULATIONAHA.106.678276. Epub 2007 Apr 23. PMID 17452608
- [Background] Yeboah J, Folsom AR, Burke GL, Johnson C, Polak JF, Post W, Lima JA, Crouse JR, Herrington DM. Predictive value of brachial flow-mediated dilation for incident cardiovascular events in a population-based study: the multi-ethnic study of atherosclerosis. Circulation. 2009 Aug 11;120(6):502-9. doi: 10.1161/CIRCULATIONAHA.109.864801. Epub 2009 Jul 27. PMID 19635967
- [Background] Gokce N, Keaney JF Jr, Hunter LM, Watkins MT, Menzoian JO, Vita JA. Risk stratification for postoperative cardiovascular events via noninvasive assessment of endothelial function: a prospective study. Circulation. 2002 Apr 2;105(13):1567-72. doi: 10.1161/01.cir.0000012543.55874.47. PMID 11927524
- [Background] Gastaldelli A, Kozakova M, Hojlund K, Flyvbjerg A, Favuzzi A, Mitrakou A, Balkau B; RISC Investigators. Fatty liver is associated with insulin resistance, risk of coronary heart disease, and early atherosclerosis in a large European population. Hepatology. 2009 May;49(5):1537-44. doi: 10.1002/hep.22845. PMID 19291789
- [Background] Villanova N, Moscatiello S, Ramilli S, Bugianesi E, Magalotti D, Vanni E, Zoli M, Marchesini G. Endothelial dysfunction and cardiovascular risk profile in nonalcoholic fatty liver disease. Hepatology. 2005 Aug;42(2):473-80. doi: 10.1002/hep.20781. PMID 15981216
- [Background] Berg AH, Scherer PE. Adipose tissue, inflammation, and cardiovascular disease. Circ Res. 2005 May 13;96(9):939-49. doi: 10.1161/01.RES.0000163635.62927.34. PMID 15890981
- [Background] Rajsheker S, Manka D, Blomkalns AL, Chatterjee TK, Stoll LL, Weintraub NL. Crosstalk between perivascular adipose tissue and blood vessels. Curr Opin Pharmacol. 2010 Apr;10(2):191-6. doi: 10.1016/j.coph.2009.11.005. Epub 2010 Jan 7. PMID 20060362
- [Background] Hopkins TA, Ouchi N, Shibata R, Walsh K. Adiponectin actions in the cardiovascular system. Cardiovasc Res. 2007 Apr 1;74(1):11-8. doi: 10.1016/j.cardiores.2006.10.009. Epub 2006 Oct 20. PMID 17140553
- [Background] Zhu W, Cheng KK, Vanhoutte PM, Lam KS, Xu A. Vascular effects of adiponectin: molecular mechanisms and potential therapeutic intervention. Clin Sci (Lond). 2008 Mar;114(5):361-74. doi: 10.1042/CS20070347. PMID 18230060
- [Background] Kaser S, Moschen A, Cayon A, Kaser A, Crespo J, Pons-Romero F, Ebenbichler CF, Patsch JR, Tilg H. Adiponectin and its receptors in non-alcoholic steatohepatitis. Gut. 2005 Jan;54(1):117-21. doi: 10.1136/gut.2003.037010. PMID 15591515
- [Background] Bonetti PO, Lerman LO, Lerman A. Endothelial dysfunction: a marker of atherosclerotic risk. Arterioscler Thromb Vasc Biol. 2003 Feb 1;23(2):168-75. doi: 10.1161/01.atv.0000051384.43104.fc. PMID 12588755